CLINICAL TRIAL: NCT05586269
Title: Intervening in Food Insecurity to Reduce and Mitigate (InFoRM) Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Allison Wu, Physician, Gastroenterology and Nutrition, Principal Investigator, Instructor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00043195
Record Dates: First submitted 2022-09-23; First posted 2022-10-19 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Obesity; Nutrition Disorders; Overnutrition, Child; Obesity
Keywords: Food Insecurity; Nutrition Security
MeSH Terms: conditions — Pediatric Obesity; Nutrition Disorders; Child Nutrition Disorders; Obesity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Dyads (caregiver + child) will be randomized to one of two intervention sequences:
  1. Meal kit intervention without delay followed by newsletter + pantry referral
  2. Newsletter + pantry referral followed by meal kit intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal Kits, Then Newsletter + Food Pantry Referral (Experimental): Dyads (caregiver + child) receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
  Interventions: Behavioral: Meal Kit Delivery; Behavioral: Newsletter + Food Pantry Referral
- Newsletter + Food Pantry Referral, Then Meal Kits (Experimental): Dyads (caregiver + child) receive a newsletter and food pantry referral. After the second study visit, they receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
  Interventions: Behavioral: Meal Kit Delivery; Behavioral: Newsletter + Food Pantry Referral

INTERVENTIONS:
Behavioral: Meal Kit Delivery — Dyads (caregiver + child) receive one meal kit delivery per week. One meal kit is designed to include two recipes and ingredients to prepare 10 servings (~2 meals for a household 5 people). Meal kits come with printed picture-based recipes in English or Spanish and access to online cooking demonstrations.
  Other Names: EatWell Meal Kits
Behavioral: Newsletter + Food Pantry Referral — Dyads (caregiver + child) receive a printed newsletter in English and Spanish that lists additional local food assistance resources. Dyads receive a referral to the clinic's associated food pantry.
  Other Names: Standard of Care

SUMMARY:
The goals of this study are to 1) pilot the feasibility of a novel meal kit delivery intervention in families and children with food insecurity and obesity and 2) evaluate the implementation of the pilot intervention.

DETAILED DESCRIPTION:
Childhood obesity prevalence is rising in the U.S. and is known to track into adulthood, increasing the risks of chronic diseases such as type 2 diabetes. Households of children with obesity also face unmet social needs, such as food insecurity. Food insecurity is associated with poorer dietary quality and higher prevalence of obesity and diabetes in adults; however, data are inconsistent and less known regarding longitudinal health effects in children. Because food insecurity and childhood obesity tend to co-occur in Black, Hispanic, and lower-income households, there is an urgent need to examine and intervene in the social determinants associated with rising childhood obesity prevalence.

ELIGIBILITY:
Child Inclusion Criteria:

* Children >=6 years and <12 years old with a BMI >=95th percentile
* Children who screen positive on the 2-item Hunger Vital Sign™
* Children living in a household of <=5 people
* Children living with an English and/or Spanish-speaking caregiver
* Children living within the EatWell delivery map boundaries in the greater Boston area

Child Exclusion Criteria:

* History of food allergies or intolerance to dairy, gluten, soy, or any potential component of the meal kit
* History of malabsorptive intestinal disease (e.g., Crohn's disease, celiac disease)
* History of type 1 or 2 diabetes
* History of solid tumor or bone marrow transplant
* Enteral tube dependence

The child's primary caregiver will be eligible for enrollment.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison J Wu, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level data may be shared upon request, under the conditions that an analysis plan is prepared and approved by the PI/Co-Is, Institutional Review Board approval has been obtained, and all necessary data sharing agreements have been executed.
Supporting Information: Study Protocol, ICF
Time Frame: Data can be requested by emailing the PI.
Access Criteria: 1. An analysis plan is prepared and approved by the PI/Co-Is,
  2. IRB approval has been obtained, and
  3. All necessary data sharing agreements have been executed.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at a primary care clinic between February and March 2023. The first participant was enrolled on February 13, 2023, and the last participant was enrolled on March 9, 2023.
Pre-assignment Details: Dyad (caregiver + child) eligibility was based child criteria and caregiver language (see Study Design). The child and their primary caregiver were enrolled in the study. There were 30 children and 29 caregivers enrolled in the study. One caregiver had two children enrolled in the study.
Groups:
- Meal Kits, Then Newsletter + Food Pantry Referral: Caregivers; Meal Kits, Then Newsletter + Food Pantry Referral: Children: Dyads (caregiver + child) receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
- Newsletter + Food Pantry Referral, Then Meal Kits: Caregivers; Newsletter + Food Pantry Referral, Then Meal Kits: Children: Dyads (caregiver + child) receive a newsletter and food pantry referral. After the second study visit, they receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
Period: First Intervention (6 Weeks)
Arm/Group | Meal Kits, Then Newsletter + Food Pantry Referral: Caregivers | Meal Kits, Then Newsletter + Food Pantry Referral: Children | Newsletter + Food Pantry Referral, Then Meal Kits: Caregivers | Newsletter + Food Pantry Referral, Then Meal Kits: Children
Started | 14 | 15 | 15 | 15
Received Intervention | 13 | 14 | 15 | 15
Completed | 10 | 11 | 12 | 12
Not Completed | 4 | 4 | 3 | 3
Not completed — Lost to Follow-up | 4 | 4 | 3 | 3
Period: Second Intervention (6 Weeks)
Arm/Group | Meal Kits, Then Newsletter + Food Pantry Referral: Caregivers | Meal Kits, Then Newsletter + Food Pantry Referral: Children | Newsletter + Food Pantry Referral, Then Meal Kits: Caregivers | Newsletter + Food Pantry Referral, Then Meal Kits: Children
Started | 10 | 11 | 12 | 12
Completed | 10 | 11 | 11 | 11
Not Completed | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Dyad (caregiver + child) eligibility was based child criteria and caregiver language (see Study Design). The child and their primary caregiver were enrolled in the study. There were 30 children and 29 caregivers enrolled in the study. One caregiver had two children enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Meal Kits, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kits | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Median (Full Range); unit: years] — Population: Caregivers and children were analyzed separately.
  years
    Child age: number analyzed (Participants) | 15 | 15 | 30
    Child age | 10 [6 to 11] | 9 [6 to 11] | 9 [6 to 11]
    Caregiver age: number analyzed (Participants) | 14 | 15 | 29
    Caregiver age | 42 [27 to 50] | 39 [31 to 50] | 42 [27 to 50]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Caregivers and children were analyzed separately. In the "Meal Kits, Then Newsletter + Food Pantry Referral" arm, one caregiver was missing information.
  Participants
    Child sex: number analyzed (Participants) | 15 | 15 | 30
    Child sex: Female | 5 | 8 | 13
    Child sex: Male | 10 | 7 | 17
    Caregiver sex: number analyzed (Participants) | 13 | 15 | 28
    Caregiver sex: Female | 12 | 13 | 25
    Caregiver sex: Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregivers and children were analyzed separately.
  Participants
    Child ethnicity: number analyzed (Participants) | 15 | 15 | 30
    Child ethnicity: Hispanic or Latino | 11 | 15 | 26
    Child ethnicity: Not Hispanic or Latino | 3 | 0 | 3
    Child ethnicity: Unknown or Not Reported | 1 | 0 | 1
    Caregiver ethnicity: number analyzed (Participants) | 14 | 15 | 29
    Caregiver ethnicity: Hispanic or Latino | 9 | 15 | 24
    Caregiver ethnicity: Not Hispanic or Latino | 4 | 0 | 4
    Caregiver ethnicity: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Caregivers and children were analyzed separately.
  Participants
    Child race: number analyzed (Participants) | 15 | 15 | 30
    Child race: American Indian or Alaska Native | 1 | 1 | 2
    Child race: Asian | 0 | 0 | 0
    Child race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Child race: Black or African American | 7 | 6 | 13
    Child race: White | 3 | 4 | 7
    Child race: More than one race | 1 | 0 | 1
    Child race: Unknown or Not Reported | 3 | 3 | 6
    Caregiver race: number analyzed (Participants) | 14 | 15 | 29
    Caregiver race: American Indian or Alaska Native | 1 | 1 | 2
    Caregiver race: Asian | 0 | 0 | 0
    Caregiver race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Caregiver race: Black or African American | 6 | 5 | 11
    Caregiver race: White | 3 | 3 | 6
    Caregiver race: More than one race | 1 | 0 | 1
    Caregiver race: Unknown or Not Reported | 3 | 5 | 8
Number of people living in the household [Median (Full Range); unit: persons] — Population: Only caregivers reported number of people living in the household. In the "Meal Kits, Then Newsletter + Food Pantry Referral" arm, one caregiver was missing information.
  persons
    Number of adults 18 years and older: number analyzed (Participants) | 13 | 15 | 28
    Number of adults 18 years and older | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
    Number of children younger than 18 years: number analyzed (Participants) | 13 | 15 | 28
    Number of children younger than 18 years | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]
Caregiver marital status [Count of Participants; unit: Participants] — Population: Only caregivers reported marital status.
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    Married | 3 | 3 | 6
    Never married | 5 | 2 | 7
    Divorced | 1 | 3 | 4
    Separated | 3 | 4 | 7
    Widowed | 1 | 0 | 1
    Prefer not to answer | 0 | 3 | 3
    Missing | 1 | 0 | 1
Total annual household income [Count of Participants; unit: Participants] — Population: Only caregivers reported household income.
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    Less than $20,000 | 7 | 10 | 17
    Between $20,000 and $70,000 | 2 | 3 | 5
    More than $70,000 | 2 | 0 | 2
    Don't know | 2 | 1 | 3
    Prefer not to answer | 0 | 1 | 1
    Missing | 1 | 0 | 1
Highest grade or degree completed [Count of Participants; unit: Participants] — Population: Only caregivers reported their highest grade or degree completed.
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    8th grade or less | 2 | 2 | 4
    Some high school | 2 | 6 | 8
    High school graduate | 3 | 4 | 7
    Some college or technical school | 2 | 1 | 3
    College graduate | 3 | 2 | 5
    Postgraduate training or degree | 1 | 0 | 1
    Don't know or prefer not to answer | 0 | 0 | 0
    Missing | 1 | 0 | 1
Caregiver relationship to child [Count of Participants; unit: Participants] — Population: Only caregivers reported their relationship to their child.
  Participants
    number analyzed (Participants) | 14 | 15 | 29
    Mother | 12 | 13 | 25
    Father | 1 | 2 | 3
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility: Recruitment
Description: Proportion of eligible participants who were recruited and enrolled in the intervention, prior to randomization.
Time Frame: 2 months to baseline
Population: All participants who met eligibility criteria after being screened.
Measure: Count of Participants; unit: Participants
Groups:
- Both Arms: The total sample is included as the proportion of eligible participants, including children and caregivers, who were recruited and enrolled in the intervention was assessed prior to randomization to one of two arms.
Arm/Group | Both Arms
Number analyzed (Participants) | 69
Participants
  Enrolled | 59
  Declined to enroll | 10

2. Primary Outcome: Study Feasibility: Randomization
Description: Number of participants enrolled per month, then subject to randomization.
Time Frame: At baseline
Population: All participants (caregivers and children) who consented to participate in the study. Randomization occurred by caregiver after completing the consent. There were 30 children and 29 caregivers enrolled in the study. One caregiver had two children enrolled in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Dyads (caregiver + child) receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
- Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Dyads (caregiver + child) receive a newsletter and food pantry referral. After the second study visit, they receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 29 | 30
Participants
  Number of participants enrolled (February) | 20 | 20
  Number of participants enrolled (March) | 9 | 10

3. Primary Outcome: Study Feasibility: Retention
Description: Number of participants retained at each study visit
Time Frame: At the baseline first study visit (baseline), at the second study visit (week 6-8), and at the third study visit (week 14-16).
Population: All participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Caregiver: Caregivers receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
- Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Children: Children receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
- Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Caregiver: Caregivers receive a newsletter and food pantry referral. After the second study visit, they receive healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
- Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Children: Children receive a newsletter and food pantry referral. After the second study visit, they receive healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Caregiver | Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Children | Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Caregiver | Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Children
Number analyzed (Participants) | 14 | 15 | 15 | 15
Participants
  First study visit: Participants remaining in study visit | 13 | 14 | 15 | 15
  First study visit: Participants lost to follow up in study visit | 1 | 1 | 0 | 0
  Second study visit: number analyzed (Participants) | 13 | 14 | 15 | 15
  Second study visit: Participants remaining in study visit | 10 | 11 | 12 | 12
  Second study visit: Participants lost to follow up in study visit | 3 | 3 | 3 | 3
  Third study visit: number analyzed (Participants) | 10 | 11 | 12 | 12
  Third study visit: Participants remaining in study visit | 10 | 11 | 11 | 11
  Third study visit: Participants lost to follow up in study visit | 0 | 0 | 1 | 1

4. Primary Outcome: Study Feasibility: Protocol
Description: Number of participants who reported receipt of all six weeks of meal kit delivery
Time Frame: Third study visit (week 14-16)
Population: All participants with assessment data at the third study visit.
Measure: Count of Participants; unit: Participants
Groups:
- Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Dyads receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
- Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Dyads receive a newsletter and food pantry referral. After the second study visit, they receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 21 | 22
Participants | 19 | 22

5. Primary Outcome: Study Feasibility: Adherence - Caregivers
Description: Total number of recipes prepared by caregivers
Time Frame: Third study visit (week 14-16)
Population: All caregivers with assessment data at the third study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 10 | 11
Participants
  Caregivers who prepared 7-12 recipes | 3 | 2
  Caregivers who prepared 3-6 recipes | 4 | 4
  Caregivers who prepared 1-2 recipes | 2 | 5
  Caregivers who did not prepare any recipe | 1 | 0

6. Primary Outcome: Study Feasibility: Adherence - Children
Description: Number of children who tasted/ate food from the meal kit
Time Frame: Third study visit (week 14-16)
Population: All caregivers with assessment data at the third study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 11 | 11
Participants | 10 | 11

7. Primary Outcome: Study Feasibility: Assessments
Description: Proportion of planned assessments completed at each study visit
Time Frame: At the baseline first study visit (baseline), at second study visit (week 6-8), and at third study visit (week 14-16)
Population: The first study visit included a baseline demographic survey, 2 child assessments, and 1 caregiver assessment. The second study visit included 2 child assessments and 1 parent assessment. The third study visit included 2 child assessments, 1 parent assessment, and 1 satisfaction questionnaire. The "Meal Kit Delivery, Then Newsletter + Food Pantry Referral" arm included 14 caregivers and 15 children (one pair of siblings), thus the discrepancy between total planned assessments in each arm.
Measure: Count of Units; unit: Survey/Assessments
Units Other Than Participants: Survey/Assessments
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 29 | 30
Number analyzed (Survey/Assessments) | 162 | 165
Survey/Assessments
  Planned assessments completed after visit 1: number analyzed (Survey/Assessments) | 59 | 60
  Planned assessments completed after visit 1 | 56 | 60
  Planned assessments completed after visit 2: number analyzed (Survey/Assessments) | 44 | 45
  Planned assessments completed after visit 2 | 32 | 35
  Planned assessments completed after visit 3: number analyzed (Survey/Assessments) | 59 | 60
  Planned assessments completed after visit 3 | 38 | 43

8. Secondary Outcome: Number of Participants With Household Food Insecurity at the First Study Visit
Description: Severity of food insecurity was assessed using the US Household Food Security Survey Module, which is categorized by the raw score into:
  Zero: High food security 1-2: Marginal food security 3-7: Low food security 8-18: Very low food security
Time Frame: At the baseline first study visit (baseline)
Population: Caregivers who reported household-level food security at baseline study visit 1 (baseline).
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 13 | 15
Participants
  High food security | 0 | 0
  Marginal food security | 1 | 0
  Low food security | 8 | 11
  Very low food security | 4 | 4

9. Secondary Outcome: Number of Participants With Household Food Insecurity at Second Study Visit
Description: as for outcome 8
Time Frame: At second study visit (week 6-8)
Population: Caregivers who reported household-level food security at study visit 2 (week 6-8).
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 10 | 12
Participants
  High | 1 | 1
  Marginal food security | 1 | 1
  Low food security | 5 | 8
  Very low food security | 3 | 2

10. Secondary Outcome: Number of Participants With Household Food Insecurity at Third Study Visit
Description: as for outcome 8
Time Frame: At third study visit (week 14-16)
Population: Caregivers who reported household-level food security at third study visit (week 14-16).
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 9 | 11
Participants
  High food security | 2 | 2
  Marginal food security | 0 | 1
  Low food security | 5 | 7
  Very low food security | 2 | 1

11. Secondary Outcome: Change in BMI For Children With BMI Assessments At All Visits
Description: Weight and height were combined to report BMI in kg/m^2 based on Centers for Disease Control growth curves.
Time Frame: At baseline, at second study visit (week 6-8), and at third study visit (week 14-16)
Population: Children with BMI data at three study visits.
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Caregivers: Caregivers receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration). After the second study visit, they receive a newsletter and food pantry referral.
- Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Caregivers: Caregivers receive a newsletter and food pantry referral. After the second study visit, they receive weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral: Caregivers | Newsletter + Food Pantry Referral, Then Meal Kit Delivery: Caregivers
Number analyzed (Participants) | 9 | 10
kg/m^2
  BMI at Baseline | 26.29 (3.07) | 24.82 (2.85)
  BMI at Visit 2 | 26.64 (2.78) | 24.67 (2.68)
  BMI at Visit 3 | 26.54 (2.81) | 24.66 (2.81)
  Change from Baseline at Visit 2 | 0.36 (1.52) | -0.15 (0.59)
  Change from Baseline at Visit 3 | 0.26 (1.77) | -0.16 (0.50)
  Change from Visit 2 and Visit 3 | -0.10 (0.62) | -0.01 (0.70)

12. Secondary Outcome: Change in BMI Percentage of the 95th Percentile for Children With BMI Assessments at All Visits
Description: BMI percentage of the 95th percentile (BMIp95) was calculated using CDC extended BMI-for-age growth charts for children with BMI assessments at all study visits
Time Frame: At baseline, at second study visit (week 6-8), and at third study visit (week 14-16)
Population: Children with BMI data at all three study visits.
Measure: Mean (Standard Deviation); unit: percentage of the 95th percentile
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 9 | 10
percentage of the 95th percentile
  BMIp95 at Baseline | 117.5 (12) | 113.3 (11)
  BMIp95 at Visit 2 | 118.5 (12) | 111.8 (12)
  BMIp95 at Visit 3 | 117.3 (12) | 111.0 (12)
  Change from Baseline at Visit 2 | 1.0 (7) | -1.5 (2)
  Change from Baseline at Visit 3 | -0.2 (8) | -2.3 (2)
  Change from Visit 2 to Visit 3 | -1.1 (3) | -0.8 (3)

13. Other Pre Specified Outcome: Total Prime Diet Quality Score at Each Study Visit: Children
Description: The PrimeScreen survey was used to assess the total prime diet quality score (PDQS) for the child (parent-reported). The survey enables calculation of a food group's daily intake frequency. Scores range from 5 (minimum) to 65 (maximum) across thirteen food groups. A higher score indicates more healthy diet quality.
Time Frame: At baseline first study visit (baseline), at second study visit (week 6-8), and at third study visit (week 14-16)
Population: Children with dietary data at study visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 14 | 15
units on a scale
  Child Prime Diet Quality Score (PDQS) at Baseline | 39 (6) | 39 (4)
  Child Prime Diet Quality Score (PDQS) at Visit 2: number analyzed (Participants) | 11 | 11
  Child Prime Diet Quality Score (PDQS) at Visit 2 | 44 (7) | 41 (4)
  Child Prime Diet Quality Score (PDQS) at Visit 3: number analyzed (Participants) | 10 | 11
  Child Prime Diet Quality Score (PDQS) at Visit 3 | 44 (7) | 43 (4)

14. Other Pre Specified Outcome: Total Prime Diet Quality Score at Each Study Visit: Caregiver
Description: The PrimeScreen survey was used to assess the total prime diet quality score (PDQS) for the caregiver (self-reported). The survey enables calculation of a food group's daily intake frequency. Scores range from 5 (minimum) to 65 (maximum) across thirteen food groups. A higher score indicates more healthy diet quality.
Time Frame: At baseline first study visit (baseline), at second study visit (week 6-8), and at third study visit (week 14-16)
Population: Parents with dietary data at study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 13 | 15
score on a scale
  Caregiver Prime Diet Quality Score (PDQS) at Baseline | 44 (6) | 42 (6)
  Caregiver Prime Diet Quality Score (PDQS) at Visit 2: number analyzed (Participants) | 10 | 12
  Caregiver Prime Diet Quality Score (PDQS) at Visit 2 | 48 (6) | 46 (5)
  Caregiver Prime Diet Quality Score (PDQS) at Visit 3: number analyzed (Participants) | 9 | 11
  Caregiver Prime Diet Quality Score (PDQS) at Visit 3 | 48 (5) | 47 (5)

15. Other Pre Specified Outcome: Caregiver Reported Mealtime Behavior at First Study Visit
Description: Caregivers rated Likert scale items from 1 (never) to 5 (everyday): "How often does your child eat dinner together with family members?"
Time Frame: At baseline first study visit (baseline)
Population: Children with parent-reported data on mealtime behavior.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 14 | 15
Participants
  Never/Less than once per week | 3 | 1
  Once per week | 0 | 1
  2-4 times per week | 5 | 2
  5-6 times per week | 1 | 1
  Everyday | 5 | 10

16. Other Pre Specified Outcome: Caregiver Reported Mealtime Behavior at Second Study Visit
Description: as for outcome 15
Time Frame: At second study visit (week 6-8)
Population: Children with parent-reported mealtime behavior data.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 11 | 12
Participants
  Never/Less than once per week | 0 | 1
  Once per week | 0 | 1
  2-4 times per week | 5 | 2
  5-6 times per week | 2 | 2
  Everyday | 4 | 6

17. Other Pre Specified Outcome: Caregiver Reported Mealtime Behavior at Third Study Visit
Description: as for outcome 15
Time Frame: At third study visit (week 14-16)
Population: Children with parent-reported mealtime behavior data.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 10 | 11
Participants
  Never/Less than once per week | 0 | 2
  Once per week | 2 | 1
  2-4 times per week | 5 | 2
  5-6 times per week | 0 | 2
  Everyday | 3 | 4

18. Other Pre Specified Outcome: Caregiver Perceived Stress at First Study Visit
Description: The Perceived Stress Scale was used to assess changes in stress (caregiver self-reported). Scores range from 0 to 40 with higher scores indicating higher perceived stress:
  0-13: low stress 14-26: moderate stress 27-40: high perceived stress
Time Frame: At baseline first study visit (baseline)
Population: Caregivers with perceived stress data.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 13 | 14
Participants
  High perceived stress | 1 | 0
  Moderate perceived stress | 7 | 7
  Low perceived stress | 5 | 7

19. Other Pre Specified Outcome: Caregiver Perceived Stress at Second Study Visit
Description: as for outcome 18
Time Frame: At second study visit (week 6-8)
Population: Caregivers with perceived stress data.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 9 | 12
Participants
  High perceived stress | 0 | 0
  Moderate perceived stress | 5 | 5
  Low perceived stress | 4 | 7

20. Other Pre Specified Outcome: Caregiver Perceived Stress at Third Study Visit
Description: as for outcome 18
Time Frame: At third study visit (week 14-16)
Population: Caregivers with perceived stress data.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Kit Delivery, Then Newsletter + Food Pantry Referral | Newsletter + Food Pantry Referral, Then Meal Kit Delivery
Number analyzed (Participants) | 8 | 11
Participants
  High perceived stress | 1 | 0
  Moderate perceived stress | 3 | 5
  Low perceived stress | 4 | 6

ADVERSE EVENTS:
Time Frame: Six weeks for each intervention.
Description: Safety Population included all participants who received at least one meal kit or the newsletter + food pantry referral.
Groups:
- Meal Kit Delivery: Caregivers: Caregivers who received weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
- Meal Kit Delivery: Children: Children who received weekly healthy meal kits with fresh ingredients and simple recipes (6 weeks duration).
- Newsletter + Food Pantry Referral: Caregivers: Caregivers who received a newsletter and food pantry referral.
- Newsletter + Food Pantry Referral: Children: Children who received a newsletter and food pantry referral.
Arm/Group | Meal Kit Delivery: Caregivers | Meal Kit Delivery: Children | Newsletter + Food Pantry Referral: Caregivers | Newsletter + Food Pantry Referral: Children
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/26

LIMITATIONS AND CAVEATS:
Consistent with the goal of the pilot phase I study, the analysis is descriptive. This phase I study was not intended to be powered to detect changes in the secondary outcomes. Secondary outcomes were collected to determine the feasibility of the assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT05586269/Prot_SAP_000.pdf